CLINICAL TRIAL: NCT00031811
Title: Breast Cancer Survivors: Exercise and Raloxifene
Brief Title: Raloxifene With or Without Exercise Compared With Exercise Alone in Women Who Have Been Previously Treated for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000069229; OHSU-6312 (Other: OHSU IRB); NCI-H02-0086
Record Dates: First submitted 2002-03-08; First posted 2003-08-06 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer; Menopausal Symptoms; Osteoporosis
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; osteoporosis; menopausal symptoms
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Raloxifene Hydrochloride

INTERVENTIONS:
Drug: raloxifene
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Raloxifene and exercise may improve bone health and quality of life in breast cancer survivors. Assessing bone health and quality of life may improve the ability to plan treatment.

PURPOSE: Randomized clinical trial to study the effectiveness of raloxifene with or without exercise compared with exercise alone in women who have been previously treated for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of raloxifene with or without exercise versus exercise alone on bone reabsorption rate, bone formation rate, and bone density in women previously treated for breast cancer.
* Determine the effects of these regimens on the quality of life of these patients.

OUTLINE: This is a randomized, placebo-controlled, multicenter study. Patients are randomized to one of four treatment arms.

* Arm I: Patients are asked to exercise 5 days a week with instruction. Patients also receive oral placebo once daily.
* Arm II: Patients receive oral raloxifene once daily.
* Arm III: Patients are asked to exercise as in arm I. Patients also receive oral raloxifene once daily.
* Arm IV: Patients receive oral placebo once daily. All patients receive oral calcium supplements once daily. Treatment continues in all arms for 24 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and every 3 months during study.

PROJECTED ACCRUAL: A total of 240 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer
* No metastatic disease
* At least 3 months but no more than 1 year since prior chemotherapy regimen including doxorubicin or methotrexate and catabolic steroids (to prevent nausea, vomiting, fluid retention, or hypersensitivity reactions)
* No routine of regular strenuous exercise (more than 90 minutes per day 6 days/week OR 120 minutes per day 4 days/week)
* Hormone receptor status:

  * Estrogen and progesterone receptor negative OR
  * Estrogen and progesterone receptor positive

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Postmenopausal (at diagnosis OR chemotherapy-induced)
* No spontaneous menses for more than 6 months with increased follicle-stimulating hormone and decreased estradiol

Performance status:

* Ambulatory

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No cardiac problems that would preclude exercise
* No unstable angina

Pulmonary:

* No respiratory problems that would preclude exercise
* No chronic obstructive pulmonary disease
* No oxygen dependence

Other:

* No endocrine disease (e.g., parathyroid hormone disorders) that would accelerate bone turnover and loss
* No musculoskeletal problems or other disease that would preclude exercise (e.g., movement-limiting arthritis, muscular dystrophy, or chronic fatigue syndrome)
* No known cognitive or psychiatric disorders that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior adjuvant or neoadjuvant chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent tamoxifen

Radiotherapy:

* Prior adjuvant radiotherapy after chemotherapy allowed
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent bisphosphonates

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-03; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schwartz, FNP, PhD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States